CLINICAL TRIAL: NCT01631201
Title: A Phase 2b, Randomized, Double-Blind, Active-Controlled Study to Evaluate the Safety and Efficacy of Rifalazil (25 Milligram) Compared With Azithromycin (1 Gram) for the Treatment of Uncomplicated Genital Chlamydia Trachomatis Infection in Women
Brief Title: Safety and Efficacy Study of Rifalazil for the Treatment of Chlamydia Trachomatis Infection in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ActivBiotics Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APL-1648-027
Record Dates: First submitted 2012-06-18; First posted 2012-06-29 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Chlamydia Trachomatis Infection
Keywords: Chlamydia
MeSH Terms: conditions — Chlamydia Infections | interventions — KRM 1648; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifalazil 25 milligram (Experimental)
  Interventions: Drug: Rifalazil 25 milligram
- Azithromycin 1 gram (Active Comparator): Single dose of Azithromycin 1 gram to be administered on Day 1.
  Interventions: Drug: Azithromycin 1 gram

INTERVENTIONS:
Drug: Rifalazil 25 milligram — Single dose of 25 milligram rifalazil to be administered on Day 1.
  Other Names: KRM-1648
  Arms: Rifalazil 25 milligram
Drug: Azithromycin 1 gram — Single dose of Azithromycin 1 gram to be administered on Day 1.
  Other Names: Zithromax
  Arms: Azithromycin 1 gram

SUMMARY:
This study will test the safety and effectiveness of an investigational antibiotic drug, rifalazil for the treatment of uncomplicated genital Chlamydia trachomatis infection. This study will examine the effects of 25 milligram of rifalazil compared with azithromycin 1 gram, which will be given as a single dose to women who have genital chlamydial infection.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 19 years old diagnosed with genital chlamydia trachomatis infection.
* Use an effective method of contraception.
* Agree to be abstinent or to have partners use condoms for all sexual activities during the study.

Exclusion Criteria:

* Subject or sexual partner is known to have gonorrhea.
* History of repeated chlamydia trachomatis infection.
* HIV, syphilis, or active Hepatitis B or C infection.
* Treatment with antimicrobial therapy with known activity against chlamydia trachomatis within 4 weeks of enrollment.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with microbiologic cure of chlamydia trachomatis infection at Day 22 | Day 22
  Microbiologic test result will be reported as positive or negative for chlamydia trachomatis.

SECONDARY OUTCOMES:
Proportion of subjects with microbiologic cure of chlamydia trachomatis infection at Day 36. | Day 36
  Microbiologic test result will be reported as positive or negative for chlamydia trachomatis.
Number of subjects experiencing adverse events in the two treatment groups. | Day 36 (end of study)
Number of subjects experiencing clinically significant laboratory abnormalities in the two treatment groups. | Day 36 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Chalom B Sayada, MD, PhD, Study Director — ActivBiotics Pharma
Locations (5):
- United States (5):
  - Research Site, Birmingham, Alabama
  - Research Site, San Diego, California
  - Research Site, Indianapolis, Indiana
  - Research Site, Las Vegas, Nevada
  - Research Site, Virginia Beach, Virginia

REFERENCES:
- [Derived] Geisler WM, Pascual ML, Mathew J, Koltun WD, Morgan F, Batteiger BE, Mayes A, Tao S, Hurwitz SJ, Sayada C, Schinazi RF. Randomized, double-blind, multicenter safety and efficacy study of rifalazil compared with azithromycin for treatment of uncomplicated genital Chlamydia trachomatis infection in women. Antimicrob Agents Chemother. 2014 Jul;58(7):4014-9. doi: 10.1128/AAC.02521-14. Epub 2014 May 5. PMID 24798277